CLINICAL TRIAL: NCT00721721
Title: Genetic Epidemiology Network of Salt Sensitivity
Brief Title: Analyzing Genetic Factors Involved in Blood Pressure Changes Due to Salt and Potassium Intake (The GenSalt Study)
Acronym: GenSalt
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Jiang He, MD, PhD, Tulane University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1412; U01HL072507 (NIH)
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-08

CONDITIONS: Blood Pressure
Keywords: Dietary Sodium; Dietary Potassium; Genes; Genomics
MeSH Terms: interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants will follow a low sodium diet for Days 1 through 7, a high sodium diet for Days 7 through 14, and a high sodium diet plus potassium supplement regimen for Days 14 through 21.
  Interventions: Behavioral: Low Sodium Diet; Behavioral: High Sodium Diet; Dietary Supplement: Potassium Supplementation

INTERVENTIONS:
Behavioral: Low Sodium Diet — 3 grams of salt or 51.3 mmol of sodium per day
Behavioral: High Sodium Diet — 18 grams of salt or 307.8 mmol of sodium per day
Dietary Supplement: Potassium Supplementation — 60 mmol potassium supplement

SUMMARY:
High blood pressure is a serious health problem. In terms of diet recommendations, people with this condition are encouraged to eat a low sodium and high potassium diet. It is believed that genetics may play a role in the development of high blood pressure and may affect changes in blood pressure levels, including changes brought on by sodium and potassium. This study will identify genetic factors that may influence blood pressure changes due to increased salt or potassium intake in people with mildly elevated blood pressure and in their family members.

DETAILED DESCRIPTION:
High blood pressure is one of the most common health problems among adults. If left untreated, it can lead to heart failure, kidney failure, or stroke. Common causes include stress, diet, diabetes, kidney disease, or obesity. Typical treatments include taking medication, losing weight, and quitting smoking. It is also recommended that people with high blood pressure or those at risk of developing high blood pressure modify their diets to decrease sodium intake and increase potassium intake. Research has shown that genetics may play a role in the development of high blood pressure and may affect fluctuations of blood pressure levels, including blood pressure changes brought on by sodium and potassium. This study will identify and analyze the genetic factors that may be responsible for blood pressure changes due to dietary salt and potassium intake. Blood samples collected in this study may also be used for future genetic research on blood pressure.

This study will enroll people who have mildly elevated blood pressure and their siblings, spouses, and children. Participants will first take part in a 3-day observation period. At a Day 1 study visit, participants' weight, height, waist size, and blood pressure will be measured. There will be three separate blood pressure measurements. Study staff will then interview participants to collect information on family and personal medical history, cigarette smoking habits, alcohol consumption, physical activity, and diet. Finally, blood samples will be collected. For 24 hours after the first study visit, participants will collect their urine. At study visits on Days 2 and 3, participants will undergo three blood pressure measurements and a cold pressor test, which measures blood pressure at different body temperatures. Participants will also collect a urine sample each night.

After the 3-day observation period, participants will take part in a 3-week treatment period. Each day, all participants will eat breakfast, lunch, and dinner in the study kitchen. For Days 1 through 7, participants will eat a low sodium diet; for Days 7 through 14, participants will eat a high sodium diet; and for Days 14 through 21, participants will eat a high sodium diet and receive potassium supplements. Blood pressure will be measured three times per day and urine will be collected at several times during this period. Blood samples will be collected at the end of each week.

Parents of participants will also be enrolled in this study, and they will complete the same study procedures that participants complete during the 3-day observation period except for the urine collection.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Primary Participants:

* Between 18 and 60 years old
* Systolic blood pressure level of 130 to 160 mm Hg and/or diastolic blood pressure level of 85 to 100 mm Hg
* Both parents (2-generation nuclear family) or at least one parent (at least a 3-generation family) is available and willing to participate in the study
* At least one sibling meets eligibility criteria for participation

Inclusion Criteria for Sibling/Spouse/Child Participants:

* Siblings and spouses must be between 18 and 60 years old; children must be more than 16 years old
* Lives in the same village as the main study participant

Exclusion Criteria for All Participants:

* Current stage 2 hypertension (systolic blood pressure level greater than or equal to 160 mm Hg and/or diastolic blood pressure level greater than or equal to 100 mm Hg)
* Current or recent (i.e., less than 1 month before the screening visit) use of antihypertensive medications or medications that affect blood pressure
* Secondary hypertension
* History of clinical cardiovascular disease, including heart attack, congestive heart failure, stroke, and peripheral arterial disease
* Chronic kidney failure or urinary albumin concentration of greater than or equal to 20 mg/dL
* Current diabetes (i.e., fasting serum glucose level greater than or equal to 126 mg/dL) or use of insulin or oral hypoglycemic agents
* Peptic ulcer disease requiring treatment in the 2 years before study entry
* Liver disease requiring treatment in the 2 years before study entry
* Pregnant
* Heavy alcohol drinker (i.e., more than 14 drinks per week)
* Currently adhering to a low sodium diet

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1906 (Actual)
Dates: Start 2003-10; Primary Completion 2005-07 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Measured at Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Jiang He, MD, PhD, Principal Investigator — Tulane University
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Result] GenSalt Collaborative Research Group. GenSalt: rationale, design, methods and baseline characteristics of study participants. J Hum Hypertens. 2007 Aug;21(8):639-46. doi: 10.1038/sj.jhh.1002207. Epub 2007 Apr 19. PMID 17443206
- [Result] Gu D, Rice T, Wang S, Yang W, Gu C, Chen CS, Hixson JE, Jaquish CE, Yao ZJ, Liu DP, Rao DC, He J. Heritability of blood pressure responses to dietary sodium and potassium intake in a Chinese population. Hypertension. 2007 Jul;50(1):116-22. doi: 10.1161/HYPERTENSIONAHA.107.088310. Epub 2007 May 7. PMID 17485599
- [Derived] Xing X, Liu F, Yang X, Huang C, Zhang D, Chen S, Chen J, Li J, Liu Z, Lu F, Gu D, Huang J. Central Blood Pressure Responses to Dietary Sodium and Potassium Interventions. Am J Hypertens. 2018 Apr 13;31(5):582-589. doi: 10.1093/ajh/hpx209. PMID 29385399
- [Derived] Gu X, Gu D, He J, Rao DC, Hixson JE, Chen J, Li J, Huang J, Wu X, Rice TK, Shimmin LC, Kelly TN. Resequencing Epithelial Sodium Channel Genes Identifies Rare Variants Associated With Blood Pressure Salt-Sensitivity: The GenSalt Study. Am J Hypertens. 2018 Jan 12;31(2):205-211. doi: 10.1093/ajh/hpx169. PMID 29036630
- [Derived] Kelly TN, Li C, Hixson JE, Gu D, Rao DC, Huang J, Rice TK, Chen J, Cao J, Li J, Anderson CE, He J. Resequencing Study Identifies Rare Renin-Angiotensin-Aldosterone System Variants Associated With Blood Pressure Salt-Sensitivity: The GenSalt Study. Am J Hypertens. 2017 May 1;30(5):495-501. doi: 10.1093/ajh/hpx004. PMID 28199472
- [Derived] Yang X, Gu D, He J, Hixson JE, Rao DC, Lu F, Mu J, Jaquish CE, Chen J, Huang J, Shimmin LC, Rice TK, Chen J, Wu X, Liu D, Kelly TN. Genome-wide linkage and regional association study of blood pressure response to the cold pressor test in Han Chinese: the genetic epidemiology network of salt sensitivity study. Circ Cardiovasc Genet. 2014 Aug;7(4):521-8. doi: 10.1161/CIRCGENETICS.113.000332. Epub 2014 Jul 15. PMID 25028485
- [Derived] Zhao Q, Gu D, Chen J, Li J, Cao J, Lu F, Guo D, Wang R, Shen J, Chen J, Chen CS, Mills KT, Schwander K, Rao DC, He J. Blood pressure responses to dietary sodium and potassium interventions and the cold pressor test: the GenSalt replication study in rural North China. Am J Hypertens. 2014 Jan;27(1):72-80. doi: 10.1093/ajh/hpt163. Epub 2013 Sep 4. PMID 24004934
- [Derived] Kelly TN, Rebholz CM, Gu D, Hixson JE, Rice TK, Cao J, Chen J, Li J, Lu F, Ma J, Mu J, Whelton PK, He J. Analysis of sex hormone genes reveals gender differences in the genetic etiology of blood pressure salt sensitivity: the GenSalt study. Am J Hypertens. 2013 Feb;26(2):191-200. doi: 10.1093/ajh/hps018. Epub 2012 Dec 28. PMID 23382403
- [Derived] Zhao Q, Gu D, Hixson JE, Liu DP, Rao DC, Jaquish CE, Kelly TN, Lu F, Ma J, Mu J, Shimmin LC, Chen J, Mei H, Hamm LL, He J; Genetic Epidemiology Network of Salt Sensitivity Collaborative Research Group. Common variants in epithelial sodium channel genes contribute to salt sensitivity of blood pressure: The GenSalt study. Circ Cardiovasc Genet. 2011 Aug 1;4(4):375-80. doi: 10.1161/CIRCGENETICS.110.958629. Epub 2011 May 11. PMID 21562341
- [Derived] Kelly TN, Hixson JE, Rao DC, Mei H, Rice TK, Jaquish CE, Shimmin LC, Schwander K, Chen CS, Liu D, Chen J, Bormans C, Shukla P, Farhana N, Stuart C, Whelton PK, He J, Gu D. Genome-wide linkage and positional candidate gene study of blood pressure response to dietary potassium intervention: the genetic epidemiology network of salt sensitivity study. Circ Cardiovasc Genet. 2010 Dec;3(6):539-47. doi: 10.1161/CIRCGENETICS.110.940635. Epub 2010 Sep 22. PMID 20861505
- [Derived] Chen J, Gu D, Huang J, Rao DC, Jaquish CE, Hixson JE, Chen CS, Chen J, Lu F, Hu D, Rice T, Kelly TN, Hamm LL, Whelton PK, He J; GenSalt Collaborative Research Group. Metabolic syndrome and salt sensitivity of blood pressure in non-diabetic people in China: a dietary intervention study. Lancet. 2009 Mar 7;373(9666):829-35. doi: 10.1016/S0140-6736(09)60144-6. Epub 2009 Feb 14. PMID 19223069